CLINICAL TRIAL: NCT00168987
Title: Pilot Study: Randomized Controlled Trial on the Influence of an Oral Nutritional Supplement Rich in Omega-3 Fatty Acids on Functional State and Quality of Life in Malnourished Patients With Gastroenterological Tumors
Brief Title: Influence of an Oral Nutritional Supplement Rich in Omega-3 Fatty Acids on Functional State and Quality of Life in Malnourished Patients With Gastroenterological Tumors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Pfrimmer Nutricia GmbH, Erlangen , Germany (Industry)
Responsible Party: Dr. Matthias Pirlich, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA1/174/05
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Colorectal Neoplasms; Hepatocellular Carcinoma; Cholangiocarcinoma
Keywords: oral nutritional supplement; eicosapentanoic acid; gastroenterological tumors; muscle function; quality of life; body composition
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Hepatocellular; Cholangiocarcinoma | interventions — Eicosapentaenoic Acid

INTERVENTIONS:
Drug: oral nutritional supplement rich in eicosapentanoic acid

SUMMARY:
Malnutrition is a frequent symptom of various malignant diseases and is frequently observed in patients with gastrointestinal tumors. Eicosapentanoic acid (EPA) has been introduced as specific and anticatabolic acting substrate in cancer patients. Only few randomized trials are available which investigated the effect of EPA in form of an EPA-enriched, protein- and energy-dense oral nutritional supplement mostly in patients with pancreatic carcinoma.

Therefore, the effect of an EPA-rich oral nutritional supplement for two months on functional state and quality of life in patients with other gastroenterological tumors and weight loss is investigated in this randomized prospective trial.

ELIGIBILITY:
Inclusion Criteria:

* malignant disease: colorectal neoplasm, hepatocellular carcinoma, cholangiocarcinoma
* palliative treatment of malignant disease: UICC stage >1
* impaired nutritional state: weight loss > 5% body weight in the preceding 6 months or subjective global assessment grade B (moderately malnourished) or grade C (severely malnourished)
* informed written consent

Exclusion Criteria:

* age < 18 years
* pregnancy
* exclusive enteral or parenteral nutrition
* taking of eicosapentanoic acid in form of fish oil capsules
* contraindications for oral nutrition (i.e. ileus, uncontrollable vomiting)
* terminal stage of disease with a life expectancy < 3 months
* missing or withdrawn consent
* simultaneous participation in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-01; Primary Completion 2006-11 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
improvement of muscle function (hand grip strength, respiratory muscle function) at two months
improvement of cognitive function at two months
improvement of quality of life at two months

SECONDARY OUTCOMES:
tolerance of the oral nutritional supplement
improvement of nutritional state (body weight, muscle mass, body cell mass, phase angle, serum albumin)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Pirlich, MD, Principal Investigator — Charite University Hospital, Dept. of Gastroenterology, Hepatology and Endocrinology
Locations (1):
- Charite University Hospital, Berlin, Germany